CLINICAL TRIAL: NCT01154504
Title: The Role of Adrenomedullin on the Outcome of Severe Heart Failure: a Clinical Randomized Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We randomized 18 patients, but was impossible to measure adrenomedullin in Brazil. However, we analysed some interesting clinical and laboratorial results.
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Anna Stein, MD, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEP1781/07
Record Dates: First submitted 2010-06-28; First posted 2010-07-01 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Heart Failure
Keywords: adrenomedullin; heart failure; ultrafiltration; hemofiltration
MeSH Terms: conditions — Heart Failure | interventions — Adrenomedullin; Ultrafiltration; Dialysis; Hemofiltration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- clinical treatment (Other): Patients with previous diagnosis of decompensated III and IV Heart Failure will be included. The clinical treatment will be optimized.
  Clinical assessment, Adrenomedullin, Angiotensin II, Brain Natriuretic Peptide, oxydative stress, sympathetic nervous system activity will be evaluated at the beginning, at discharge and 90 days after randomization(plus or minus3).
  Interventions: Other: clinical treatment
- ultrafiltration (Experimental): ultrafiltration will be done on decompensated patients III and IV acute heart failure on Intensive Care Unit. This patients will have biochemical analysis, adrenomedullin, angiotensin II,Brain Natriuretic Peptide, oxydative stress measurements,sympathetic nervous system activity evaluated and clinical outcome analyzed at the beginning,at discharge and 90 days after randomization(plus or minus 3).
  Diuretic will be withdrawn during ultrafiltration.
  Interventions: Procedure: ultrafiltration
- isovolumetric hemofiltration (Experimental): Patients randomized to this group will have isovolumetric hemofiltration on Intensive Care Unit. They will have biochemical analysis, Adrenomedullin plasmatic level, Brain Natriuretic Peptide Level, Angiotensin II level, Oxydative stress measurement,sympathetic nervous system, and clinical outcome evaluated at the study beginning,at discharge and 90 days after randomization(plus or minus 3).
  Interventions: Procedure: isovolumetric hemofiltration

INTERVENTIONS:
Other: clinical treatment — The clinical treatment will be optimized to gold standard international heart failure treatment
  Other Names: adrenomedullin
  Arms: clinical treatment
Procedure: ultrafiltration — The ultrafiltration procedure will be done on Intensive Care Unit with automatic machine and HF 1400 filter. The fluid will be removed until a increased of 10% in hematocrit or clinical improvement.
  Other Names: dialysis; adrenomedullin
  Arms: ultrafiltration
Procedure: isovolumetric hemofiltration — The isovolumetric hemofiltration will be done in Intensive Care Unit for 8 hours, and will be permitted the diuretic use.The dose will be 35 ml/kg/hour and will e used automatic machine and MF1400 filter.Diuretic use will be maintained.
  Other Names: hemofiltration; dialysis; adrenomedullin
  Arms: isovolumetric hemofiltration

SUMMARY:
1. Study Hypothesis:

   * The decrease of plasma adrenomedullin (ADM) concentration by ultrafiltration and isovolumetric hemofiltration in patients with acute III and IV Class New York Heart Association Functional(NYHA) heart failure is more pronounced than a standard diuretic treatment and is related with clinical improvement.
2. Outcome Measurements:

To correlate the adrenomedullin plasma levels with clinical treatment, ultrafiltration and hemofiltration related to:

* Brain natriuretic peptide (BNP) level
* angiotensin II level
* sympathetic nervous activity
* oxydative stress
* clinical outcome at the beginning, at discharge and 90 days after randomization.

DETAILED DESCRIPTION:
Testing the hypothesis that adrenomedullin (ADM) is a important peptide in severe heart failure and that is related to clinical condition, we will study the effects of 3 different treatments (clinical usual treatment,ultrafiltration and isovolumetric hemofiltration with diuretics) to participants are followed until discharge to Adrenomedullin level and clinical outcomes,and also their relationship with angiotensin II level, brain natriuretic peptide(BNP), sympathetic nervous system and oxydative stress.

The patients will be randomized in three different treatment group and analyzed in three moments: on the randomization, at discharge and 90 days after randomization(plus or minus 3).

The clinical treatment will be optimized, the ultrafiltration will be done until clinically adequate fluid removal or until hematocrit increased 10% from basal level, and isovolumetric hemofiltration will be done for 8 hours- dose of 35 ml/kg/h in association with diuretic. All this dialytic procedures will be done with PAES membrane- filter HF1400 and automatic machine.

ELIGIBILITY:
Inclusion Criteria:

* more than two item:

  * more than eighteen years of age
  * orthopnea
  * Chest Rx with cardiomegaly and pulmonary infiltration
  * edema
  * diuretic resistance

Exclusion Criteria:

* insulin dependent diabetes
* hepatic cirrhosis
* vascular access problems
* creatinine more than 2,5 mg/dl before acute heart failure
* systemic infection
* aortic stenosis and heart transplantation
* radiologic contrast up to 72 hours prior randomization
* advanced neoplasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Levels of Adrenomedullin plasma in different treatments- clinical,ultrafiltration and isovolumetric hemofiltration | 90 days after randomization (plus or minus 3 days).
  The adrenomedullin level will be compared in three different treatments: clinical treatment, ultrafiltration treatment and isovolumetric hemofiltration.
Levels of Adrenomedullin plasma in different treatments- clinical,ultrafiltration and isovolumetric hemofiltration | at discharge
  The adrenomedullin level will be compared in three different treatments: clinical treatment, ultrafiltration treatment and isovolumetric hemofiltration. The patients will be followed until discharge.

SECONDARY OUTCOMES:
The Adrenomedullin plasma levels in three different treatment approaches will be related to clinical outcome. | at discharge
  The correlation of adrenomedullin plasma levels in all 3 arms related to optimized clinical outcome. The patients will be followed until discharge
The Adrenomedullin plasma levels in three different treatment approaches will be related to clinical outcome. | 90 days after randomization (plus or minus 3)
  The correlation of adrenomedullin plasma levels in all 3 arms related to optimized clinical outcome.
The Adrenomedullin plasma levels in three different treatment approaches will be related to oxydative stress | at discharge
  The correlation of adrenomedullin plasma levels in all 3 arms related to oxydative stress. The patients will be followed until discharge.
The Adrenomedullin plasma levels in three different treatment approaches will be related to oxydative stress | 90 days after randomization(plus or minus 3)
  The correlation of adrenomedullin plasma levels in all 3 arms related to oxydative stress.
The Adrenomedullin plasma levels in three different treatment approaches will be related to angiotensin II plasma level | at discharge
  The correlation of adrenomedullin plasma levels in all 3 arms related to angiotensin II level. The patients will be followed until discharge.
The Adrenomedullin plasma levels in three different treatment approaches will be related to angiotensin II plasma level | 90 days after randomization(plus or minus 3)
  The correlation of adrenomedullin plasma levels in all 3 arms related to angiotensin II plasma level.
The Adrenomedullin plasma levels in three different treatment approaches will be related to Brain natriuretic peptide plasma level | at discharge
  The correlation of adrenomedullin plasma levels in all 3 arms related to Brain natriuretic peptide level. The patients will be followed until discharge.
The Adrenomedullin plasma levels in three different treatment approaches will be related to Pro-Brain natriuretic peptide plasma level | 90 days after randomization(plus or minus 3)
  The correlation of adrenomedullin plasma levels in all 3 arms related to Brain natriuretic peptide level, 90 days after randomization(plus or minus 3)
The Adrenomedullin plasma levels in three different treatment approaches will be related to sympathetic nervous system activity | at discharge
  The correlation of adrenomedullin plasma levels in all 3 arms related to sympathetic nervous system.The patients will be followed until discharge.
The Adrenomedullin plasma levels in three different treatment approaches will be related to sympathetic nervous system activity | 90 days after randomization(plus or minus 3)
  The correlation of adrenomedullin plasma levels in all 3 arms related to sympathetic nervous system.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Cardiologia, Porto Alegre, Rio Grande do Sul, Brazil